CLINICAL TRIAL: NCT00148070
Title: Phase II Study of Tailored-Dose Docetaxel in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Rhone-Poulenc Rorer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 9900; GIA#11119; IRBMED 1999-121
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Docetaxel — You will then receive your first dose of docetaxel chemotherapy. It is put through your IV over 1-2 hours. you will receive docetaxel every 3 weeks in the Cancer Center Infusion area.
Procedure: Erythromycin Breath Test (ERMBT) — you will have an erythromycin breath test, which is an experimental test which is used to estimate the amount of enzyme produced by your liver which can metabolize the chemotherapy, docetaxel. For this test, you go to the GCRC where you will receive an injection of erythromycin (an antibiotic) which is labeled with a very small amount of radioactive substance. 20 minutes later you will blow air from your mouth into a blue solution until it clears. Your doctors will calculate the dose of docetaxel to be given to you based on this blood test, on your body's albumin level (a protein determined on the blood test), and on your height and weight.

SUMMARY:
This is a research study which aims to improve the way that doctors determine the dose of chemotherapy given to patients. Right now, chemotherapy is determined by a patient's height and weight. However, some patients metabolize chemotherapy faster or slower than the average person because of a different level of drug metabolizing enzyme in the liver. Therefore, some patients are either given too small or too large a dose of chemotherapy because the amount of enzyme is not taken into account. This research study will examine the use of a simple test, call the Erythromycin Breath Test(ERMBT) to determine the amount of enzyme which can metabolize the chemotherapy drug docetaxel (Taxotere). The dose of docetaxel will be tailored to the amount of enzyme which is available to metabolize the drug for each patient.

DETAILED DESCRIPTION:
This is a research study which aims to improve the way that doctors determine the dose of chemotherapy given to patients. Right now, chemotherapy is determined by a patient's height and weight. However, some patients metabolize chemotherapy faster or slower than the average person because of a different level of drug metabolizing enzyme in the liver. Therefore, some patients are either given too small or too large a dose of chemotherapy because the amount of enzyme is not taken into account. This research study will examine the use of a simple test, call the Erythromycin Breath Test(ERMBT) to determine the amount of enzyme which can metabolize the chemotherapy drug docetaxel (Taxotere). The dose of docetaxel will be tailored to the amount of enzyme which is available to metabolize the drug for each patient. Patients participating in this study will have biopsy proven, measurable metastatic breast cancer.

During the study:

-Patients will receive tailored-dose docetaxel for their breast cancer.

Approximately 45 subjects will be recruited at this site.

Diagnosis and Staging

•All patients will have primary tumor measurements by physical exam and/or radiographic studies (CT, MRI, bone scan).

Erythromycin Breath Test* •The ERMBT will be administered in the outpatient setting, prior to the first cycle of docetaxel. Twenty minutes after the injection of a trace amount of (14C N-methyl) erythromycin, (This test assesses the activity of the cytochrome P450 enzyme which is largely responsible for the metabolism of the chemotherapeutic agent docetaxel.)patients will exhale through a tube creating bubbles in a solution of hyamine hydroxide, ethanol, and a blue indicator until 2 mmol of carbon dioxide has been trapped and the blue color vanishes.

Premedications

* Dexamethasone 8 mg po bid for three days, beginning the day prior to docetaxel administration.
* Diphenhydramine 50 mg IVPB
* Granisetron 2 mg po 30 minutes pre-docetaxel

Chemotherapy

* Docetaxel, tailored dose, to be infused over 1 hour on day 1 every 3 weeks for the duration of study.
* Starting dose of docetaxel to be determined by the ERMBT and serum albumin according to formula as stated in protocol (page 11).

Suggested post-chemotherapy antiemetics:

•Compazine 10 mg po q 6 hours prn nausea/vomiting

Pharmacokinetic Analysis

•All patients will have pharmacokinetic determination with blood drawn for pharmacokinetic analysis over a 24 hour period after the first docetaxel treatment. Time points include time 0, 15 minutes, 45 minutes, 180 minutes (3 hours), 390 minutes (6.5 hours), and 1440 minutes (24 hours).

DEXA Scan*

* DEXA scan will be performed during the patient's stay in the Clinical Research Center, on the Lunar DPXL Bone Densitometer. This is a very simple and noninvasive test which uses x-rays and a computer program to analyze the ratio of 38 keV to 70 keV attenuation. The program then calculates Fat and Lean values for the arms, legs, abdomen, ribs, and the total body. This is the same test that is in widespread clinical use for the evaluation of osteoporosis. During the DEXA scan, patients will be exposed to a trace amount of radiation which is equal to about 2% of the yearly background dose, or less.

  *The amount of radiation to be administered by the erythromycin breath test and DEXA scan is not medically significant.
* After the first dose of docetaxel, patients will receive docetaxel every 3 weeks

How long a patient continues on chemotherapy will be decided by both the patient and the doctor. If a patient is responding to docetaxel, typically they receive 6-8 doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven, measurable metastatic breast cancer. Patients with bone-only, and/or effusion-only disease are excluded.
* Karnofsky performance status equal to 70 or greater.
* ANC > 1500, Hgb > 10, plt > 100.
* Patients with some degree of hepatic dysfunction and renal dysfunction are encouraged, in order to evaluate the ability of the ERMBT in tailoring dose in these patient populations.

Exclusion Criteria:

* Age less than 18 years.
* Allergy to erythromycin.
* Previous treatment with docetaxel. Prior paclitaxel is allowed.
* Grade > 2 peripheral neuropathy.
* No confounding factors present to provide misinterpretation of data (i.e., concurrent malignancy).
* Patients who are pregnant or nursing will not be eligible for this protocol. Women of childbearing age who are not practicing reliable birth control must have a documented negative serum HCG.
* Patients who require concurrent treatment with drugs which are known to induce or inhibit CYP3A activity will be ineligible for the trial. This list includes the drugs midazolam, anti-mycotic agents (ketoconazole and related compounds), macrolide antibiotics (erythromycin and related compounds), nifedipine, anti-seizure drugs, and rifampin (induction).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 1999-03; Primary Completion 2004-09 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To assess whether assignment of docetaxel dose based on the ERMBT will result in decreased variability in drug area under the curve when compared to dosing based on body surface area. | 12 months

SECONDARY OUTCOMES:
To evaluate the safety and efficacy of tailored-dose docetaxel in metastatic breast cancer. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Schott, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States